CLINICAL TRIAL: NCT05922683
Title: Ability of the Probiotic Vivomixx to Improve Environmental Enteropathy in Pregnant Women: a Proof of Concept Trial in Bangladesh, Pakistan, Senegal, and Zambia
Brief Title: Maternal Probiotic Intervention to Improve Gut Health
Acronym: MPIGH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); International Centre for Diarrhoeal Disease Research, Bangladesh (Other); University of Zambia (Other); Institut Pasteur de Dakar (Other)
Responsible Party: Principal Investigator, Dr Syed Asad Ali, professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 51975
Record Dates: First submitted 2023-06-20; First posted 2023-06-28 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Environmental Enteric Dysfunction; Stunting
Keywords: probiotic; microbiome; pregnant women; capscan device; urine LR; vivomixx; pakistan; malnourished children; biomarkers; EED
MeSH Terms: conditions — Growth Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomisation will be carried out using sealed envelopes, using a randomisation code prepared by the trial statistician, which will be stratified by study centre. Each woman who gives consent will be given a trial identification (TID) number which will match the number on the randomisation envelopes.
  The trial will be blinded with an identical placebo (microcrystalline cellulose, prepared by Mendes SA, Lugano). Samples will be run and analysed using TID only, with all data cleaning and re-assays carried out blinded. The trial statistician will unblind lab data once databases are finalised.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vivomixx (Experimental): Participant in the treatment arm will receive a daily dose of the probiotic Vivomixx for 8 weeks.
  Interventions: Drug: Vivomixx; Device: CapScan®
- Placebo (Placebo Comparator): Participant in the control arm will receive a daily dose of a placebo (microcrystalline maltose) for 8 weeks.
  Interventions: Device: CapScan®

INTERVENTIONS:
Drug: Vivomixx — Vivomixx (a mixture of Lactobacillus acidophilus, Lactobacillus plantarum, Lactobacillus casei, Lactobacillus delbrueckii subspecies bulgaricus, Streptococcus salivarius subspecies thermophiles, Bifidobacterium breve, Bifidobacterium longum, and Bifidobacterium infantis), as VivomixxAll consenting participants will be randomized into the treatment to control arm, receiving either Vivomixx or a placebo for 8 weeks.
  During the study, women will visit the healthcare center or vice-versa on a bi-weekly basis to receive sachets of Vivomixx or a placebo according to their trial arm.
  Other Names: VSL#3
  Arms: Vivomixx
Device: CapScan® — The only non-standard sample collection instrument is the CapScan device. The CapScan Collection Capsule ("Capsule") is a non-invasive device that collects gastrointestinal samples along the GI tract that are then analyzed outside the body. Samples collected by the Capsule will be expressed, then undergo DNA sequencing and mass spectrometric analysis to determine the identity and function of the bacterial and host cells in the different regions of the GI tract and compared to similar analyses conducted on concomitantly collected stool samples.

SUMMARY:
There is an urgent need to identify interventions that can improve the supportive uterine environment in which the fetus establishes his/her growth. Investigators believe that this necessitates improving the delivery of nutrients to the mother, and in turn that requires a healthy microbiota. Reducing intestinal inflammation will also have a profound impact on maternal and fetal immunity, though there is limited information on the impact of maternal health on placental function. This trial will determine if a well-established probiotic, Vivomixx, can modulate the maternal microbiota and ameliorate the maternal environmental enteropathy which compromises growth in the first 1000 days. This trial is the first in a proposed series of proof-of-concept intervention studies that are intended to provide data to enable a rational selection of interventions to be evaluated at scale in future large-scale trials.

This initial study will also serve the purpose of developing a harmonized multi-site Experimental Medicine Platform across four countries (Bangladesh, Pakistan, Senegal, Zambia). Harmonized procedures will develop the capacity to deliver high-quality trials for the evaluation of potential interventions to improve maternal nutritional status and growth in utero. To this end, measuring and understanding variability in endpoint measurements is a key deliverable.

DETAILED DESCRIPTION:
76 healthy pregnant women in their second trimester will be enrolled and will be randomized to receive either probiotic or placebo for 8 weeks. It will be a double-blind trial.

Pregnant women will be recruited in the community through demographic surveillance system established in Matiari, Pakistan. The study staff will approach the potential participants and will introduce them to this study. If Participants agree, a screening consent form will be taken in which investigators will assess them clinically and will measure their hemoglobin level and gestational ultrasound for confirmation of their trimester/gestational weeks. Based on the screening results and clinical staff assessment, women will be enrolled after taking trial participation consent.

Once the participant is enrolled, investigators will collect blood, urine LR, and stool samples (flash frozen and CapScan) before giving either a placebo or probiotic(which will be replenished after every 3 days). investigators will then follow them weekly for compliance and adverse event data collection for 56 days (8 weeks). investigators will again collect the same blood and stool samples after completion of 56 days. An additional visit at 36 weeks will be done to record weight and for a gestational ultrasound. Pregnancy outcomes will be recorded and then the child will be followed at 3,6,9 and 12 weeks for anthropometry and morbidity data collection. Gestational ultrasounds will be performed at screening at 20, 28 and 36 weeks of gestation.

ELIGIBILITY:
Inclusion Criteria:

* Women over the age of 18 in their second trimester of pregnancy living in defined geographical areas of Matiari, where it can be assumed that environmental enteropathy is universal.

Exclusion Criteria:

* have had diarrhoea, defined as the passage of three or more loose stools per 24 hours, in the preceding 14 days;
* have taken antibiotics or probiotics in the preceding 14 days;
* have taken non-steroidal anti-inflammatory drugs or steroids in the preceding 14 days;
* have haemoglobin concentration <8g/dl;
* have any illness which in the opinion of the investigator will complicate assessment of safety or efficacy;
* have any gastrointestinal contraindication to ingestion of a capsule (known or suspected gastrointestinal obstruction, stricture, fistula, gastroparesis, or any swallowing disorder);
* have a plan to leave the study area within the follow-up period;

but may be enrolled if/when these disqualifiers have expired.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 76 (Actual)
Dates: Start 2023-08-09 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Reduction in inflammation and epithelial damage in pregnant women with environmental enteropathy | Day 0 (screening) - Day 56
  Percentage change (mean, unweighted) in a multiple panels of biomarkers between baseline and last sample collected after 56 days of treatment, compared to a control group.

SECONDARY OUTCOMES:
Reduction in enteropathogen colonisation | Day 1 - Day 56
  Reduction in colonisation with specific enteropathogens (Salmonella, Shigella, Campylobacter, ETEC, EPEC, EAEC, rotavirus, norovirus, Giardia and Cryptosporidium), by qPCR, between baseline and last sample collected after 56 days of treatment, in Vivomixx compared to placebo groups
Impact of Vivomixx on the structure and function of the microbiome | Day 1 - Day 56
  Change in relative abundance values of alpha and beta diversity pre- and post-treatment samples.
Vivomixx Reduction in permeability | Day 1 - Day 56
  Reduction in LR ratio in Vivomixx compared to placebo groups
Impact of the host metabolome in pregnant woman | Day 1 - Day 56
  Change in the metabolome, Untargeted urine, and plasma (and fecal) metabolome before and after the intervention.
Rate of weight gain in the 2nd trimester of pregnancy | Day 1 - Day 56
  Weight gain velocity in the 2nd trimester of pregnancy
Variability in endpoints across geographies and participating laboratories | Day 1 - Day 56
  Measurements of variability, including standard deviations and kappa values; Preliminary work across all sites using identical kits and harmonised SOPs

OTHER OUTCOMES:
CapScan success rate in delivering an assessment of the microbiome throughout the gut | Day 1 - Day 56
  Recovery of useful data from CapScan; completion of whole gut microbiome profiles
Impact on growth of the infant | Day 189 - Day 554
  Growth of infant during first year by measuring WHZ score on quarterly basis
Impact of Vivomixx on intra-uterine growth restriction velocity | Day 1 - 161 Days
  Ultrasound evaluation of intrauterine growth.

CONTACTS AND LOCATIONS:
Overall Officials: Asad Ali, MPH, Principal Investigator — Aga Khan University Hospital, Karachi
Locations (1):
- Mother and Child Health Research and Training Center, Matiari, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available within 24 months of study completion.
Access Criteria: Data access requests will be reviewed by the Trial Management Group. Requestors will be required to sign a Data Access Agreement.